# Informed Consent Form – Parent

21.03.2024

### Royal Brompton Hospital



#### **Patient Identification Number for this study:**

#### **INFORMED CONSENT FORM**

**Title:** The ACTIVELY study - Evaluation of exercise testing and physical activity in children and adolescents living with inherited arrhythmias

Name of Researcher: Catherine Renwick

| | Please |
|---|---|
| | initial box |
| <ol> <li>I confirm that I have read and understand the information sheet dated 24<sup>th</sup> April<br/>2024 (Version 1.0) for the above study and have had the opportunity to consider<br/>the information, ask questions and have these answered satisfactorily.</li> </ol> | |
| 2. I was developed the transport wild/s provide action in such patents and the success for a term | 1 |
| <ol> <li>I understand that my child's participation is voluntary, and they are free to<br/>withdraw at any time, without giving any reason, without medical care or legal<br/>rights being affected.</li> </ol> | |
| | 1 |
| 3. I understand that relevant sections of any of my child's medical notes and data collected during the study may be looked at by responsible individuals from the study Sponsor or from regulatory authorities where it is relevant to my child taking part in research. I give permission to these individuals to have access to my child's records. | |
| 4. The same of the three models and the same three Cabbs about the same disable and the | T |
| 4. I agree with the publication of the results of this study in a medical journal (all data will be published anonymously). | |
| <ol><li>I agree to /my child's GP being informed about /my child's participation in this<br/>study.</li></ol> | |
| | 1 |
| 6. I agree to my child taking part in the above study. | |
| 7. My child has any known allergies to ECG stickers. | |
| Please provide details so alternative options for ECG stickers can be provided | |
| 8. I would like to be kept informed of the study's results. | |
| Please provide email contact details | |

## Royal Brompton Hospital



| Name of Child | Date | Signature |
|-------------------------------|------|-----------|
| Name of Parent | Date | Signature |
| Name of person taking consent | Date | Signature |

When completed 1 for patient; 1 for researcher; 1 (original) to be kept with hospital notes